CLINICAL TRIAL: NCT05117489
Title: A Phase 1b, Open-Label Study Evaluating the Safety, Efficacy, and Pharmacokinetics of Miricorilant in Adult Patients With Presumed Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Study Evaluating the Safety, Efficacy, and Pharmacokinetics of Miricorilant in Patients With Presumed Nonalcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CORT118335-861
Record Dates: First submitted 2021-10-12; First posted 2021-11-11 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
Keywords: Nonalcoholic Steatohepatitis; NASH; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — CORT118335

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Cohort 1 - 150 mg of miricorilant for 24 weeks (Experimental): Patients who meet the entry criteria for study CORT-118335-861 will be enrolled to receive miricorilant as a steady dose of 150 mg once daily, for 24 weeks.
  Interventions: Drug: Miricorilant 150 mg
- Cohort 2 - 150 mg of miricorilant for 12 weeks (Experimental): Patients who meet the entry criteria for study CORT-118335-861 will be enrolled to receive miricorilant as a steady dose of 150 mg once daily, for 12 weeks.
  Interventions: Drug: Miricorilant 150 mg
- Cohort 3 - 100 mg daily miricorilant for 2 weeks, followed by 100 mg every MWF for 10 weeks (Experimental): Patients who meet the entry criteria for study CORT-118335-861 will be enrolled to receive miricorilant as a steady dose of 100 mg once daily for 2 weeks, followed by 100 mg of miricorilant every Monday, Wednesday and Friday for 10 weeks.
  Interventions: Drug: Miricorilant 100 mg
- Cohort 4 - 100 mg daily miricorilant for 2 weeks, followed by 100 mg every MF for 10 weeks (Experimental): Patients who meet the entry criteria for study CORT-118335-861 will be enrolled to receive miricorilant as a steady dose of 100 mg once daily, for 2 weeks, followed by 100 mg of miricorilant every Monday and Friday for 10 weeks.
  Interventions: Drug: Miricorilant 100 mg
- Cohort 5 - 100 mg of miricorilant every MWF for 12 weeks (Experimental): Patients who meet the entry criteria for study CORT-118335-861 will be enrolled to receive miricorilant of 100 mg every Monday, Wednesday and Friday for 12 weeks.
  Interventions: Drug: Miricorilant 100 mg
- Cohort 6 - 100 mg of miricorilant every MF for 12 weeks (Experimental): Patients who meet the entry criteria for study CORT-118335-861 will be enrolled to receive miricorilant of 100 mg every Monday and Friday for 12 weeks.
  Interventions: Drug: Miricorilant 100 mg
- Cohort 7 - 50 mg of miricorilant daily for 12 weeks (Experimental): Patients who meet the entry criteria for study CORT-118335-861 will be enrolled to receive miricorilant as a steady dose of 50 mg once daily, for 12 weeks.
  Interventions: Drug: Miricorilant 50 mg
- Cohort 8 - 100 mg of miricorilant daily for 12 weeks (Experimental): Patients who meet the entry criteria for study CORT-118335-861 will be enrolled to receive miricorilant as a steady dose of 100 mg once daily, for 12 weeks.
  Interventions: Drug: Miricorilant 50 mg
- Cohort 9 - 30 mg of miricorilant daily for 12 weeks (Experimental): Patients who meet the entry criteria for study CORT-118335-861 will be enrolled to receive miricorilant as a steady dose of 30 mg once daily, for 12 weeks.
  Interventions: Drug: Miricorilant 10 mg
- Cohort 10 - 200 mg of miricorilant once a week for 12 weeks (Experimental): Patients who meet the entry criteria for study CORT-118335-861 will be enrolled to receive miricorilant as a steady dose of 200 mg once weekly, for 12 weeks.
  Interventions: Drug: Miricorilant 50 mg
- Cohort 11 - 150 mg of miricorilant twice weekly for 12 weeks (Experimental): Patients who meet the entry criteria for study CORT-118335-861 will be enrolled to receive miricorilant as a steady dose of 150 mg twice weekly for 12 weeks.
  Interventions: Drug: Miricorilant 50 mg

INTERVENTIONS:
Drug: Miricorilant 150 mg — Miricorilant 150 mg for oral dosing
  Other Names: CORT118335
  Arms: Cohort 1 - 150 mg of miricorilant for 24 weeks; Cohort 2 - 150 mg of miricorilant for 12 weeks
Drug: Miricorilant 100 mg — Miricorilant 100 mg for oral dosing
  Other Names: CORT118335
  Arms: Cohort 3 - 100 mg daily miricorilant for 2 weeks, followed by 100 mg every MWF for 10 weeks; Cohort 4 - 100 mg daily miricorilant for 2 weeks, followed by 100 mg every MF for 10 weeks; Cohort 5 - 100 mg of miricorilant every MWF for 12 weeks; Cohort 6 - 100 mg of miricorilant every MF for 12 weeks
Drug: Miricorilant 50 mg — Miricorilant 50 mg for oral dosing
  Other Names: CORT118335
  Arms: Cohort 10 - 200 mg of miricorilant once a week for 12 weeks; Cohort 11 - 150 mg of miricorilant twice weekly for 12 weeks; Cohort 7 - 50 mg of miricorilant daily for 12 weeks; Cohort 8 - 100 mg of miricorilant daily for 12 weeks
Drug: Miricorilant 10 mg — Miricorilant 10 mg for oral dosing.
  Other Names: CORT118335
  Arms: Cohort 9 - 30 mg of miricorilant daily for 12 weeks

SUMMARY:
This phase 1b, Open-Label Study is to assess the safety, efficacy of miricorilant in patients with presumed Nonalcoholic Steatohepatitis (NASH)

DETAILED DESCRIPTION:
This phase 1b, Open-Label Study will assess the safety, efficacy and pharmacokinetics (PK) of miricorilant in patients with presumed Nonalcoholic Steatohepatitis (NASH).

Patients who meet the criteria for the study CORT-118335-861 will be enrolled on Day 1 into 1 of 11 cohorts and receive:

* Cohort 1 - a daily dose of 150 mg of miricorilant over 24 weeks.
* Cohort 2 - a daily dose of 150 mg of miricorilant over 12 weeks.
* Cohort 3 - a daily dose of 100 mg of miricorilant over 2 weeks, followed by 10 weeks of dosing at 100 mg miricorilant every Monday, Wednesday and Friday.
* Cohort 4 - a daily dose of 100 mg of miricorilant over 2 weeks, followed by 10 weeks of dosing at 100 mg miricorilant every Monday and Friday.
* Cohort 5 - a thrice weekly dose of 100 mg of miricorilant over 12 weeks every Monday, Wednesday, and Friday.
* Cohort 6 - a twice weekly dose of 100 mg of miricorilant over 12 weeks every Monday and Friday.
* Cohort 7 - a daily dose of 50 mg of miricorilant over 12 weeks.
* Cohort 8 - a daily dose of 100 mg of miricorilant over 12 weeks.
* Cohort 9 - a daily dose of 30 mg of miricorilant over 12 weeks.
* Cohort 10 - a once weekly dose of 200 mg of miricorilant over 12 weeks.
* Cohort 11 - a twice weekly dose of 150 mg miricorilant over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Have a diagnosis of NASH based on a biopsy obtained within the last year OR Have a diagnosis of presumed NASH based on blood tests and scans

Exclusion Criteria:

* Have participated in another clinical trial within the last year and received active treatment for NASH
* Have participated in another clinical trial for any other indication within the last 3 months
* Are pregnant or lactating women
* Have a BMI <18 kg/m2
* Have had liver transplantation or plan to have liver transplantation during the study
* Have type 1 diabetes or poorly controlled type 2 diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Relative change from Baseline in liver-fat content assessed by MRI-PDFF compared to Baseline. | Baseline Day 1 up to Week 24

SECONDARY OUTCOMES:
Change from Baseline in aspartate aminotransferase (AST). | Baseline Day 1 up to Week 24
Change from Baseline in alanine aminotransferase (ALT). | Baseline Day 1 up to Week 24
Change from Baseline in gamma-glutamyl transferase (GGT). | Baseline Day 1 up to Week 24
Change from baseline in enhanced liver fibrosis score (ELF). | Baseline Day 1 up to Week 24
  ELF numerical values are calculated from serum measurements of hyaluronic acid (HA), tissue inhibitor of metalloproteinases-1 (TIMP-1), and type III procollagen (PIIINP) using the formula: ELF score = 2.494 + 0.846 In [HA] + 0.735 In [PIIINP] + 0.391 In [TIMP-1], and range on a continuous scale. Liver fibrosis is unlikely with scores <6.7 and increasingly likely with higher scores.

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Juneja, MD, Study Director — Corcept Therapeutics
Locations (9):
- United States (9):
  - Site 207, Chandler, Arizona
  - Site 209, Tucson, Arizona
  - Site 214, Panorama City, California
  - Site 233, Santa Ana, California
  - Site 211, Austin, Texas
  - Site 213, Edinburg, Texas
  - Site 305, Houston, Texas
  - Site 212, San Antonio, Texas
  - 226, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No